CLINICAL TRIAL: NCT04872647
Title: Pilot of Virtual Health Coaching Utilizing Lifestyle for Under-Resourced Patients With Type II Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beacon Health System (Other)
Collaborators: Beacon Health Foundation (Unknown); Coach Me Health (Unknown)
Responsible Party: Principal Investigator, Kimberly R Azelton, Family Medicine Physician, Health Services Management Fellow, Beacon Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2127
Record Dates: First submitted 2021-04-14; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Type2 Diabetes
Keywords: Socio economic status; Health Coaching; Lifestyle Medicine; Underserved

STUDY DESIGN:
Intervention Model Description: Pilot Randomized Control Trial comparing usual diabetic care to usual diabetic care plus virtual health coaching utilizing lifestyle action plans in under resourced adults with type II diabetics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Diabetic Care (No Intervention): Usual diabetic care for this study will include a diabetic visit with their primary care provider at the beginning and end of the 12 weeks. They will also be asked to continue their current level of physical activity and eating habits.
- Usual Diabetic Care Plus Virtual Health Coaching (Experimental): For the duration of the 12 weeks, Healthy at Home will provide health coaching in 10-20 minute phone calls weekly. They will request daily blood glucose logs as this is part of Healthy at Home's normal procedure. The health coach and subject will choose a patient-directed overarching goal such as "lose weight," or improve my blood sugar numbers," etc. that the health coach will then help the patient turn into a SMART goal. They will do this by utilizing a list of lifestyle change categories as top priority goals from which to choose from in their patient-directed health coaching sessions. Texting will be utilized to request daily blood glucose and provide real-time coaching via text.
  Interventions: Behavioral: Phone-Based Health Coaching Utilizing Lifestyle Action Plans

INTERVENTIONS:
Behavioral: Phone-Based Health Coaching Utilizing Lifestyle Action Plans — Culturally sensitive health coaches trained in motivational interviewing provide 10-20 minutes of weekly phone-based health coaching. They not only guide the patient in creating a SMART goal, but assess and build off of the previous weeks' goal and problem-solve with the patient. During the week, the coach and patient text regarding daily blood glucose monitoring with real-time feedback and coaching about the implementation of the patients' goal.
  Arms: Usual Diabetic Care Plus Virtual Health Coaching

SUMMARY:
Accessible and effective interventions for chronic diseases such as diabetes are especially needed in the under-resourced patient population. This is a pilot randomized control trial compares usual diabetic care to usual diabetic care plus virtual health coaching utilizing lifestyle action plans in under-resourced adult type II diabetic patients. This is a one-site study at an under-resourced family medicine residency clinic. The primary outcome is the change of insulin resistance as measured by HOMA2-IR. Secondary metabolic outcomes are being tracked. Potentially confounding variables related to SDoH, race, and engagement in health coaching are being assessed for. The cost of the intervention as well as expensive healthcare utilization as measured by ER visits are also being tracked.

DETAILED DESCRIPTION:
Those having difficulty with SDoH (Social Determinants of Health) are associated with a higher incidence of diabetes as well as worse health outcomes. Inexpensive, effective virtual options for chronic diseases conducive to all levels of socio-economic status would be very beneficial. As early as 1934 there have been reports of nutritional interventions preventing and reversing DMII. A recent randomised trial utilizing meal replacement and caloric restriction noted greater diabetes remission rates with greater weight loss. Despite knowledge that weight and dietary factors are at the foundation of DMII incidence, control and even remission, it is challenging to find accessible, effective, community-based interventions.

Culturally sensitive health coaches trained to use motivational interviewing to create specific, measurable, attainable, reasonable and time-bound (S.M.A.R.T.) action plans through shared-decision making and thus personalized to the patients' literacy, resources and motivation level may overcome some of these cultural and literacy barriers. Accessibility is further increased by utilizing phone and text. This allows for low-tech, inexpensive remote patient monitoring. This real-time feedback may further increase patient self-efficacy and engagement. While using health coaching methods may improve diabetic control, the exact content of what should be delivered is unexplored. The mixed results of diabetes remission rates in dietary intervention studies is attributed to delivery of too low a "therapeutic dose" of lifestyle change. Therefore, it is postulated that health coaches personalizing the behavioral interventions that may be most effective in controlling and reversing diabetes may improve insulin resistance in a real-world primary-care based setting to those most challenged by barriers to care.

This is a pilot randomized control trial comparing usual care to usual care plus virtual health coaching utilizing lifestyle action plans in adult type II diabetic patients. This is a one-site study at an under-resourced family medicine residency clinic. The primary outcome is the change of insulin resistance as measured by HOMA2-IR. Secondary metabolic outcomes are being tracked. Potentially confounding variables related to SDoH, race, and engagement in health coaching are being assessed for. The cost of the intervention as well as expensive healthcare utilization as measured by ER visits are also being tracked.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes (Hemoglobin A1C 6.5% or higher in the last year) who are regular patients of E. Blair Warner Clinic. English or Spanish speaking patients will be included who are between 18 and 65 years old with a working phone. Subjects recently started on or taking a short dose of medications that are known to influence insulin resistance (i.e. atypical antipsychotics, steroids, thiazides). Subjects (and their providers) on chronic doses of these medications will be asked to keep the dose the same.

Exclusion Criteria:

* Patients whose preferred language is not English or Spanish will be excluded due to lack of health coaches speaking other languages. Approximately 50% of C-peptide is cleared by the kidney and some studies excluded advanced renal failure. For our study subjects with chronic renal failure with a GFR <45 on most recent blood work will be excluded. Subjects with conditions known to influence insulin resistance (i.e. pregnancy, hemochromatosis, polytransfused individuals) will be excluded. Subjects with syndromic obesity (i.e. hypothalamic obesity, pradi-willi syndrome) or type I diabetes mellitus will be excluded. Subjects with diagnosed diseases that would hinder giving consent or participating in health coaching (i.e. dementia, cognitive impairment) will be excluded. Subjects who have attended an intensive lifestyle change program and/or made an impacting lifestyle change in the last 3 months, such as losing 5% or more of their body weight in the last 3 months will also be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-05-20 (Estimated); Study Completion 2021-05-20 (Estimated)

PRIMARY OUTCOMES:
Change of HOMA2-IR | Beginning and End of 12 Weeks
  Homeostatic Model Assessment of Insulin Resistance as a surrogate measure of upstream diabetic control

SECONDARY OUTCOMES:
sBP | Beginning and End of 12 Weeks
  systolic blood pressure in mm Hg
dBP | Beginning and End of 12 Weeks
  diastolic blood pressure in mm Hg
BMI | Beginning and End of 12 Weeks
  Body Mass Index as an aggregate of weight and height
Hemoglobin A1C | Beginning and End of 12 Weeks
  Measure of downstream diabetic control
Change in Diabetic Medications | Beginning and End of 12 Weeks
  change in number of the diabetic medications at the beginning and end of the 12 weeks
EVS | Beginning and End of 12 Weeks
  Exercise Vital Sign: minutes of exercise per day * days per week

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly R Azelton, MD, Principal Investigator — Beacon Health System; Karin Underwood, MBA, Study Chair — Coach Me Health
Locations (1):
- Beacon Health System, South Bend, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
IPD sharing would be considered on a case-by-case basis while in communication with Beacon IRB.

REFERENCES:
- [Background] Himsworth HP. Dietetic factors influencing the glucose tolerance and the activity of insulin. J Physiol. 1934 Mar 29;81(1):29-48. doi: 10.1113/jphysiol.1934.sp003113. No abstract available. PMID 16994524
- [Result] Goel A. In type 2 diabetes, a primary care-led weight management program increased weight loss and diabetes remission at 2 years. Ann Intern Med. 2019 Aug 20;171(4):JC17. doi: 10.7326/ACPJ201908200-017. No abstract available. PMID 31426060
- [Result] Walker RJ, Strom Williams J, Egede LE. Influence of Race, Ethnicity and Social Determinants of Health on Diabetes Outcomes. Am J Med Sci. 2016 Apr;351(4):366-73. doi: 10.1016/j.amjms.2016.01.008. PMID 27079342
- [Derived] Azelton KR, Crowley AP, Vence N, Underwood K, Morris G, Kelly J, Landry MJ. Digital Health Coaching for Type 2 Diabetes: Randomized Controlled Trial of Healthy at Home. Front Digit Health. 2021 Nov 25;3:764735. doi: 10.3389/fdgth.2021.764735. eCollection 2021. PMID 34901926